CLINICAL TRIAL: NCT05337215
Title: The Effect of Postpartum Kangaroo Father Care on Paternal Attachment: A Randomized Controlled Study Turkey Sample
Brief Title: The Effect of Postpartum Kangaroo Father Care on Paternal Attachment
Acronym: kangaroocare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator, Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HititUniversity_2
Record Dates: First submitted 2022-03-28; First posted 2022-04-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nursing Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): While the IIF was applied to control group at the first meeting in the postpartum ward, FIAS was administered by phone or home visit in the third month after the face-to-face interview.There was any intervention for this group
  Interventions: Behavioral: kangaroo father care
- kangaroo father care (Experimental): While the IIF was applied to control group at the first meeting in the postpartum ward, FIAS was administered by phone or home visit in the third month after the face-to-face interview.. the first KC was applied within the first 4-6 hours after birth, and the second KC was applied in the postpartum ward under the supervision of the researcher on the first day after birth. The third KC was performed by the fathers themselves at home on the third postpartum day after discharge. Immediately afterwards, the researcher observed the father and baby from an appropriate distance, and the father and the baby had skin-to-skin contact for mean 15-20 minutes.
  Interventions: Behavioral: kangaroo father care

INTERVENTIONS:
Behavioral: kangaroo father care — The effect of postpartum kangaroo father care on paternal attachment

SUMMARY:
Objective: This study was conducted in a randomized controlled manner to determine the effect of kangaroo care (KC) on paternal attachment (PA).

DETAILED DESCRIPTION:
Objective: This study was conducted in a randomized controlled manner to determine the effect of kangaroo care (KC) on paternal attachment (PA).

Design: The data for the study were collected using the introductory information form (IIF) and the father-infant attachment scale (FIAS). T test, Mann Whitney U test and Kruskal Wallis test were used for statistical analysis.

Participants and setting: A total of 90 fathers, including 45 in the intervention group and 45 in the control group who met the inclusion criteria of the study were included randomly.

Keywords: Kangaroo care; father; paternal attachment; Turkey.

ELIGIBILITY:
Inclusion Criteria:

* fathers who are aged 18 and 50,
* married,
* voluntarily agree to participate in the study,
* have healthy babies,
* live with their babies.

Exclusion Criteria:

* a history of chronic psychiatric illness
* antipsychotic medication use
* babies with premature / low birth weight / congenital anomalies

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Father-Baby Attachment Scale The Turkish version | 12 months
  Father-Baby Attachment Scale The Turkish version was applied by Güleç and Kavlak (2013) to the fathers of infants aged 6-12 months, and the McDonald coefficient was reported to be between 0.52 and 0.80 (Güleç and Kavlak 2013). The scale consists of 19 items and three sub-dimensions: "patience and tolerance". "pleasure in interaction", and "love and pride". Each item on the scale is scored between 1 and 5 points. The minimum score that can be obtained from the scale is 19 and the maximum is 95. High scores indicate that the attachment level is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Yıldırım, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No